CLINICAL TRIAL: NCT06923566
Title: Targeted Muscle Reinnervation in the Hand for the Managment of Symptomatic Neuroma Following Digit and Hand Amputations, A Prospective Case Series
Brief Title: Targeted Muscle Reinnervation in the Hand for the Managment of Symptomatic Neuroma Following Digit and Hand Amputations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 145/2021
Record Dates: First submitted 2025-03-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-03

CONDITIONS: Targeted Muscle Reinervation; Digital Amputation; Neuroma
Keywords: Targeted muscle reinnervation; neuroma; amputation
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- targeted muscle reinervation post digit amputation group (Experimental): In 1ry TMR ,after the amputation is performed by the standard method , transected nerves will be replanted micro surgically to motor entry points (MEPS)in the hand as predetermined by Daugherty et al , Motor branches in the recipient muscles could be determined by a nerve stimulator intraoperatively.
  In 2ry TMR , neuroma site will be explored and it will be excised ,the distal end of the transected nerve will be connected micro surgically to the nearest MEPS
  Interventions: Procedure: Targeted muscle reinnervation

INTERVENTIONS:
Procedure: Targeted muscle reinnervation — In 1ry TMR ,after the amputation is performed by the standard method , transected nerves will be replanted micro surgically to motor entry points (MEPS)in the hand as predetermined by Daugherty et al , Motor branches in the recipient muscles could be determined by a nerve stimulator intraoperatively.
  In 2ry TMR , neuroma site will be explored and it will be excised ,the distal end of the transected nerve will be connected micro surgically to the nearest MEPS

SUMMARY:
Neuromas are a common complication after digital and hand amputations, resulting in significant pain, discomfort, and functional impairment. Various management methods are available, including surgical excision, nerve blocks, and nerve stump protectors, but these treatments may have limited success rates and potential complications. Targeted muscle reinnervation (TMR) is a promising technique that involves surgically rerouting a severed nerve into a nearby muscle, which can prevent the formation of neuromas and provide improved muscle function

ELIGIBILITY:
Inclusion Criteria:

* Arabic or English speaking individuals
* An upper limb amputation distal to the wrist crease
* A symptomatic neuroma within the hand or digits: defined as patient-reported localized pain consistent with a clinical exam of a neuroma pain.There must be a supporting Tinel's sign on physical exam.

Exclusion Criteria:

* Cognitive impairment for better assessment of patient reported outcomes and filling questionnaires and signing consents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Neuroma incidence | through study completion, an average of 1 year
  Neuroma incidence post TMR operation is recorded via Tinel's sign
Neuroma recurrence | through study completion, an average of 1 year
  Neuroma recurrence in cases of 2ry TMR cases
Pain intensity | will be taken at intervals over time (1 month, 3 months,6 months, 9 months,1 year until the conclusion of the study
  measured using pain rating numerical scale commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable
Pain medication usage type | Followed up at intervals over time (1 month, 3 months,6 months, 9 months,1 year until the conclusion of the study
  pain medication usage type recorded
Pain medication usage frequency | Followed up at intervals over time (1 month, 3 months,6 months, 9 months,1 year until the conclusion of the study
  pain medication usage frequency recorded
Pain character | will be taken at intervals over time (1 month, 3 months,6 months, 9 months,1 year until the conclusion of the study
  Leeds Assessment of neuropathic symptoms and signs pain scale is a valuable tool designed to evaluate and categorize pain. Its primary purpose is to determine if nerve damage is the primary cause of the pain, distinguishing between neuropathic and nociceptive pain.
  The scale comprises seven items, divided into two sections. The first part consists of five questions related to symptoms experienced by the individual. The second part involves two clinical examination items that are typically conducted in collaboration with a healthcare provider.
  A score of 12 or more on this scale confirms a diagnosis of neuropathic pain to some degree. Scores below 12 are less likely to show neuropathic pain
Pain character | will be taken at intervals over time (1 month, 3 months,6 months, 9 months,1 year until the conclusion of the study
  The McGill Pain Questionnaire is a well-known assessment tool used to quantify and understand the subjective experience of pain. It primarily consists of three major categories of word descriptors-sensory affective, and evaluative-through which patients can express and specify their pain experience. In addition to these descriptors, the questionnaire includes an intensity scale and other items to further capture the properties of the pain being experienced.

SECONDARY OUTCOMES:
operative time | intraoperative
  measuring the operative time
Rate of infection | up to 30 days postoperative
  surgical site infections were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Ibrahim Fathy Aly Howeidy, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University Faculty of medicine, Al ‘Abbāsīyah, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No